CLINICAL TRIAL: NCT00005794
Title: A Phase I Trial of Perifosine on a Loading Dose/Maintenance Dose Schedule in Patients With Advanced Cancer
Brief Title: Perifosine in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 1999-355; P30CA014520 (NIH); WCCC-CO-99906; ASTA-D-21266; NCI-T99-0036; CDR0000067752 (Other: UWCCC? Unknown)
Record Dates: First submitted 2000-06-02; First posted 2003-10-08 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2015-10

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — perifosine

INTERVENTIONS:
Drug: perifosine

SUMMARY:
RATIONALE: Perifosine may stop the growth of tumor cells by stopping blood flow to the tumor.

PURPOSE: Phase I trial to study the effectiveness of perifosine in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose (MTD) of perifosine on a loading dose/maintenance dose schedule in patients with advanced solid tumors.
* Determine the qualitative and quantitative toxic effects of this drug in these patients.
* Determine the pharmacokinetics of this drug in these patients.
* Investigate the relationship between pharmacokinetic parameters and toxicity of this drug in these patients.
* Determine the recommended starting dose for phase II trials on this drug schedule in these patients.
* Evaluate the pharmacodynamic parameters on peripheral blood lymphocytes both before and during drug administration in these patients.
* Determine any changes in the MTD with prolonged administration (3 months, 6 months) of this drug in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive a loading dose of oral perifosine 4 times a day for 4-8 doses followed by a daily maintenance dose. Treatment continues every 28 days in the absence of unacceptable toxicity or disease progression.

Cohorts of 3-6 patients receive escalating loading doses and maintenance doses of perifosine until the maximum tolerated dose (MTD) of each is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxic effects.

PROJECTED ACCRUAL: Approximately 20-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed locally unresectable or metastatic malignancy that is considered incurable
* Refractory to further treatment with known forms of effective therapy
* No clinically active CNS metastasis

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* WBC at least 4,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin normal
* SGOT no greater than 2.5 times upper limit of normal

Renal:

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 6 months after study participation
* Maintaining a reasonable state of nutrition consistent with weight maintenance

  * No recent history of weight loss greater than 10% of current body weight
* No frequent vomiting/poor alimentation
* No other serious concurrent medical illness that would preclude study therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunotherapy

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for mitomycin and nitrosoureas) and recovered
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy

  * Patients who have progressive disease while being treated with LHRH agonists, antiestrogens, or antitestosterones for at least 3 months may remain on these agents if in their best interest

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* At least 21 days since prior major surgery

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-02; Study Completion 2003-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Van Ummersen, MD, Study Chair — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin, United States